CLINICAL TRIAL: NCT01595607
Title: The Influence of Daily Consumption of Avocado on Biomarkers of Vascular Health
Brief Title: The Effect of Avocado Consumption on Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS39
Record Dates: First submitted 2012-02-07; First posted 2012-05-10 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Focus: Avocado Consumption & Vascular Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Typical American Diet (Active Comparator): Participants will receive a typical American diet for 6 weeks.
  Interventions: Other: Diet Treatment
- Avocado Diet (Experimental): Participants will receive a modified typical American diet in which avocado is substituted for foods that contain moderate and high amounts of saturated fat to allow the inclusion of avocado.
  Interventions: Other: Diet Treatment

INTERVENTIONS:
Other: Diet Treatment — Participants will consume a controlled diet for 6 weeks where all meals will be provided by the facility. Participants will be instructed to eat all foods and only foods provided to them.

SUMMARY:
The study will investigate the effect of avocado consumption on markers of vascular health. Sixty participants will be enrolled in the 6-week study. A randomized parallel design will be utilized. Participants will either receive a typical American diet, or a modified typical American diet in which avocado is substituted for foods that contain moderate and high amounts of saturated fat, to allow the isoenergetic inclusion of avocado.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 42 kg/m2
* Age 28 to 70 years during the intervention
* Fasting glucose ≤ 126 mg/dl
* Blood pressure ≤ 160/100 mm Hg

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases, or malabsorption syndromes
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who routinely participate in "heavy" exercise or volunteers who initiate an exercise program during the study.
* Volunteers who have lost 10% of body weight within the last 12 months
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanalamine, ephedrine, caffeine, during and for at least 6 months prior to the start of the study) or history of a surgical intervention for obesity
* Active cardiovascular disease (such as heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months)
* Smokers or other tobacco users (during the 6 months prior to the start of the study)
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion.)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Function | 0 hr and 3 hr at baseline and after 6 weeks
  Noninvasive endothelial function will be assessed, following a 12-hours fast, by measuring endothelium-dependent flow mediated dilation of the peripheral bed. Participants will then consume a test meal and endothelial function will be assessed again 3 hours later.

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline and after 6 weeks
  Blood pressure will be measured using a standardized protocol at the beginning and end of the intervention.
Change in Gene Expression | Baseline and after 6 weeks
  Blood samples will be used to test how the intervention affects gene expression. The expression of genes related to cardiovascular disease risk will be measured at the beginning and end of the 6-week intervention (fasted and post-prandially).
Change in Biomarkers of Cardiovascular Disease Risk | Baseline and after 6 weeks
  Blood will be collected at the beginning and end of the dietary intervention, following the endothelial function measurements (fasted and post-prandial collections). Blood will be assessed for biomarkers of cardiovascular disease risk, including electrolytes (sodium, potassium, chloride), markers of inflammation (IL-6, IL-10, IL-1 beta, C-reactive protein, TNF-alpha, fibrinogen, ICAM), markers of vascular function (endothelin-1, factor VII, plasminogen), and blood lipid panel (plasma total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides).

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States